CLINICAL TRIAL: NCT04553315
Title: The Effect of Chest Expansion Exercises on Reducing Pulmonary Infection and Complications in Patients With Pleural Effusion
Brief Title: the Effect of Chest Expansion Exercises on Pleural Effusion
Acronym: PE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sarah Asmaa (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, Sarah Asmaa, clinical professor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Chest expansion exercises; sasmaa (Registry Identifier: assiut university)
Record Dates: First submitted 2020-08-30; First posted 2020-09-17 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Pulmonary Infection; Complication
Keywords: Chest expansion exercises; complications; pleural effusion; pulmonary infection
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Intervention Model Description: implementing chest expansion exercises on patient with pleural effusion to evaluate its efficacy on preventing pulmonary infection and complications
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Intervention group was received Chest mobility exercises with Incentive spirometer and segmental breathing exercise and breath stacking technique . The patient in the intervention group was instructed to perform the exercises 3 times per day, 7-8 times per session for one week. Ensure that the patient fully hydrated by maintaining normal daily water requirement in the form of (30-35ml/kg/day) with restriction of intravenous fluids.
  Interventions: Procedure: chest expansion exercises
- control group (Experimental): control group will receive only routine hospital care
  Interventions: Procedure: chest expansion exercises

INTERVENTIONS:
Procedure: chest expansion exercises — Chest mobility exercises with Incentive spirometer and segmental breathing exercise ) and breath stacking technique e.

SUMMARY:
the study attempted to assess and evaluate the efficacy of implementing chest expansion exercises on patients with pleural effusion and how this programme contribute to reduce pulmonary infection and complications.

To address the objective of the study, the researcher utilized chest expansion exercises consisted of stacked breathing exercise, segmental breathing, chest mobility exercises, deep breathing exercise with use of incentve spirometer and assess the patient before and after exercises by using three tools help to monitor hemodynamic parameters, chest condition, laboratory investigations which help to evaluate pulmonary infection score and complications.

DETAILED DESCRIPTION:
Introduction Plural effusion is a syndrome occurs frequently in hospitalized patients, leading to increased morbidity, mortality, and healthcare expenditure. A plural effusion represents the disturbance of the normal mechanisms of formation and drainage of fluid from the plural space .

Plural effusion is defined as a ﬂuid collection between the plural leaves due to local/systemic disease of the pleura, lung or extra-pulmonary organs. Normally, 0.1 to 0.2 ml/kg of ﬂuid is present in the plural leaves to facilitate plural movement. When the balance between the production and re-absorption of this ﬂuid deteriorates, it becomes plural effusion .

The accumulation of plural effusion has important effects on respiratory system function. It changes the elastic equilibrium volumes of the lung and chest wall, resulting in a restrictive ventilatory effect, chest wall expansion and reduced efficiency of the inspiratory muscles. The magnitude of these alterations depends on the plural fluid volume and the underlying disease of the respiratory system. The decrease in lung volume is associated with hypoxemia mainly due to an increase in right to left shunt. The drainage of pleural fluid results in an increase in lung volume that is considerably less than the amount of aspirated fluid, while hypoxemia is not readily reversible upon fluid aspiration .

Pleural effusions are traditionally classified as either transudates or exudates. Diseases that affect the filtration of pleural fluid result in transudate formation and often occur bilaterally. Inflammation or injury increases pleural capillary membrane permeability to proteins and various types of cells and lead to the formation of an exudative effusion .

This study was designed as a randomised controlled trial to determine the effect of chest expansion exercises on reducing pulmonary infection and complications on patients with plural effusion.

Methods Design Structured as a randomized-controlled prospective study, the objective of this study was to determine the efficacy of the chest expansion exercises on reducing pulmonary infection and complications on patients with plural effusion.

Setting Data was collected from chest ICU and critical ICU in Assiut university hospital .

Sample The study population consisted of patients eighteen to sixty years old, hospitalized and treated in Critical, Chest intensive care units. The inclusion criteria stipulated that the patient was between eighteen and sixty years old; both genders were included; diagnosed as plural effusion by the physician; and with a symmetrical chest expansion and agreed to participate in the study. A power calculation estimated that in order to detect an effect size of 0.29 difference in mean of pulmonary function between the two studied groups, with a p-value < 0.05 and 80 % power, confidence level 0.95, a sample size of 20 patients for each group was needed. However, 60 patients were attempted in this research work to avoid non-response rate (30 for each group). This calculated using G Power 3.1 . The study data was collected between June 2019 and June 2020.

Instruments and measurements Three tools used in this study were developed by the researcher based on reviewing of the relevant literature.

The first tool was Plural effusion assessment sheet used to monitor hemodynamic parameters included (Mean arterial pressure (MAP) taken from bed side monitor, heart rate (HR), temperature, respiratory rate and CVP readings, assessment of respiratory system consisted of : Chest examination done every shift before and after exercise, chest x-ray assessment, Sputum and blood culture assessment, Ventilator profile assessment , assessment of plural procedures done, assessment of clinical pulmonary infection score, fluid balance assessment., assessment of laboratory findings in addition to socio-demographic and medical data.

The second tool is Chest expansion exercises sheet : was developed by the researcher and used to assess exercises done to the patient and included: Chest mobility exercise; Stacked breathing exercise; Segmental breathing exercise; Deep breathing exercise and Incentive spirometer exercise.

The third tool is Patients' outcomes evaluation sheet which was developed by the researcher and used to assess the effect of chest expansion exercises on pulmonary infection score and complications.

Intervention After getting ethical clearance patients were enrolled in the study, patients were selected based on the inclusion and exclusion criteria. Following an initial assessment, the patients were assigned to one of the two groups by block randomization.

Intervention group was received Chest mobility exercises with Incentive spirometer and segmental breathing exercise and breath stacking technique . The patient in the intervention group was instructed to perform the exercises 3 times per day, 7-8 times per session for one week. Ensure that the patient fully hydrated by maintaining normal daily water requirement in the form of (30-35 ml/kg/day) with restriction of intravenous fluids.

Data collection The data were collected from the first day of admission after stabilization of the patient's condition and extended to 7 days, every day and every shift then the data were recorded in the developed tools.The researcher assigned study sample (30 patients) to two groups (Control group, Intervention group).

For the control group: The researcher assessed patients who were receiving the routine hospital care. For Intervention group: The researcher assessed patients then applying chest expansion exercises.

Ethical considerations There was no risk for study subject during application of the study as the study followed common ethical principles in clinical research and has been carried out in accordance with The Code of Ethics of the World Medical Association (Declaration of Helsinki) and written consent was obtained from patients or guidance that participated in the study after explaining the nature and purpose of the study.

Patient was assured that the data of this research was not be reused without second permission, confidentiality and anonymity was assured and the patients had the right to refuse to participate or withdraw from the study without any rational at any time.

Data analysis Data were computerized and analyzed by computer programmed SPSS (ver.16). Data were presented by using descriptive statistics in the form of frequencies and percentages or means ± standard deviations for qualitative data. Quantitative data were compared using Independent samples t-test for comparisons among two groups. Qualitative variables were compared using chi-square test to determine significance. The critical value of the tests "P" was considered statistically significant when P less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 - 60 years.
2. patients of both genders.
3. patients diagnosed as pleural effusion by the physician.
4. patients with asymmetrical chest expansion.

Exclusion Criteria:

1. Orthopedic conditions.
2. Pleural effusion due to transudate conditions like: liver cirrhosis, …. etc.
3. Malignant conditions.
4. Cognitive impairments.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
score of pulmonary infection | 1 year
  through the study pulmonary infection will be assessed by using pulmonary infection score by assessing parameters as WBCs, temperature and chest condition
rate of complications | 1 year
  complications will be assessed through the study by using evaluation outcomes tool

CONTACTS AND LOCATIONS:
Overall Officials: Amal A Mohamed, Principal Investigator — Assiut University
Locations (1):
- Faculty of Nursing, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD